CLINICAL TRIAL: NCT05733455
Title: Insulin Resistance in the Pathogenesis of Non-Alcoholic Fatty Liver Disease: Alpelisib Pilot & Feasibility Study
Brief Title: Effect of Alpelisib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AAAU3423
Record Dates: First submitted 2023-02-03; First posted 2023-02-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Insulin Resistance; Hyperinsulinemia; Dyslipidemias
Keywords: Insulin resistance; Hyperinsulinemia; Diabetes; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism; Dyslipidemias; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — Alpelisib; microcrystalline cellulose; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Alpelisib treatment (Experimental): Participants will ingest a single dose of alpelisib 300 mg (two overencapsulated 150-mg tablets)
  Interventions: Drug: Alpelisib 150 mg [Piqray], 2 overencapsulated tablets (total: 300 mg); Device: FreeStyle Libre Pro; Diagnostic Test: Oral glucose tolerance test (OGTT) with Trutol glucose beverage; Dietary Supplement: BOOST Plus nutritional beverage
- Placebo treatment (Placebo Comparator): Participants will ingest a single dose of placebo (two capsules filled with microcrystalline cellulose)
  Interventions: Drug: Placebo (microcrystalline cellulose), 2 capsules; Device: FreeStyle Libre Pro; Diagnostic Test: Oral glucose tolerance test (OGTT) with Trutol glucose beverage; Dietary Supplement: BOOST Plus nutritional beverage

INTERVENTIONS:
Drug: Alpelisib 150 mg [Piqray], 2 overencapsulated tablets (total: 300 mg) — Participants will ingest two overencapsulated tablets of alpelisib at 23:00, along with a saltine cracker.
  Other Names: Piqray
  Arms: Alpelisib treatment
Drug: Placebo (microcrystalline cellulose), 2 capsules — Participants will ingest two capsules filled with microcrystalline cellulose at 23:00, along with a saltine cracker.
  Arms: Placebo treatment
Device: FreeStyle Libre Pro — Continuous glucose monitoring for 24 hours (double blinded)
Diagnostic Test: Oral glucose tolerance test (OGTT) with Trutol glucose beverage — Participants will drink Trutol glucose beverage (D-glucose 75 g in 10 fl oz) and blood will be sampled at baseline and at 15, 30, 60, 90, 120, 150, and 180 minutes.
Dietary Supplement: BOOST Plus nutritional beverage — Participants will consume a quantity of BOOST Plus calculated to match their daily caloric needs, divided over three liquid meals.

SUMMARY:
The goal of this clinical trial is to test a single dose of the phosphoinositide-3-kinase (PI3K) inhibitor alpelisib versus placebo in healthy volunteers. The main questions it aims to answer are the impact of acute alpelisib-induced insulin resistance on parameters of glucose and lipid metabolism (how healthy people respond to temporary insulin resistance so that the investigators can see what happens to how the liver handles fat and sugar).

Participants will:

* Consume their total calculated daily caloric needs in nutritional supplements, divided in three meals, and otherwise fast for 24 hours
* Take a dose of alpelisib 300 mg or placebo at bedtime
* Wear a continuous glucose monitor for 72 hours
* Participate in an oral glucose tolerance test (OGTT)

Researchers will compare blood tests before and during OGTT in participants randomized (like the flip of a coin) to alpelisib versus placebo to see how the drug treatment affects plasma glucose, serum insulin, and serum lipid parameters (triglycerides, free fatty acids, and apolipoprotein B).

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an under-appreciated complication of lipid dysmetabolism in type 2 diabetes (T2DM). Although it appears that insulin resistance (IR) is a mechanism common to both, the mechanisms linking IR to unhealthy fat accumulation in liver remains unclear. "Pure" IR would be expected to disinhibit hepatic glucose production while dampening hepatic triglyceride (TG) biosynthesis, but the excessive hepatic de novo lipogenesis (DNL) of IR-associated NAFLD (IR-NAFLD) suggests that hepatic IR is "selective." However, the concept of IR selectivity is controversial, and because of clinical heterogeneity, lead-time discrepancies, co-morbidities, and medication effects, parsing out this pathophysiologic conundrum in humans is challenging. The investigators ultimately plan to test whether the multifactorial IR in patients with NAFLD is selective by determining if inducing a discrete, "pure" form of IR, via pharmacologic inhibition of phosphoinositide-3-kinase (PI3K) with alpelisib, attenuates excessive DNL. However, because of the potential toxicities of alpelisib, the investigators first must test whether they can induce IR with a single dose. In order to ensure participants' safety, the investigators propose herein to perform a randomized, placebo-controlled, pilot & feasibility study of a single dose of alpelisib in healthy volunteers. Following a baseline blood draw on Day 1, participants will be fitted with a continuous glucose monitor. Once lab test results are confirmed as non-exclusionary, randomized participants will be instructed on Day 3 to consume their calculated total daily caloric needs in the form of a nutritional beverage, divided evenly over three meals, and otherwise will fast. On the evening of Day 3, participants will ingest a single dose either of placebo or alpelisib. The following morning (Day 4), about 10 hours later, blood will be drawn to check fasting levels of glucose, insulin, and certain lipid/lipoprotein parameters; the continuous glucose monitor will be removed at that point. Participants will then undergo an oral glucose tolerance test (OGTT) during which investigators will measure glucose, insulin, and lipid (triglycerides, free fatty acids) levels. If the investigators are able to determine reliable induction after a single dose of alpelisib, they will be able to move on to test its effect on volunteers with IR-NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years, using highly effective contraception if of childbearing potential
2. Able to understand written and spoken English and/or Spanish
3. Body mass index of 18.0-26.9 kg/m2
4. Healthy, as determined by screening assessments and Principal Investigator's (PI's) clinical/scientific judgment. "Healthy" status is defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead EKG, and laboratory tests on blood and urine.

Exclusion Criteria:

1. Inability to provide informed consent in English or Spanish
2. Concerns arising at screening visit (any of the following):

   i. Unwillingness to fast (except water) for up to 15 hours

   ii. Documented weight change of ≥ 3.0% of baseline within the previous 6 months

   iii. Abnormal blood pressure
   * Systolic blood pressure < 90 mm Hg or > 160 mm Hg, and/or
   * Diastolic blood pressure < 60 mm Hg or > 100 mm Hg

   iv. Abnormal resting heart rate ≤ 60 bpm or ≥ 100 bpm
   * Sinus tachycardia that has been extensively worked up and considered benign by the recruit's personal physician may be permitted at the PI's discretion

     v. Abnormal screening electrocardiogram (or if on file, performed within previous 90 d)
   * Non-sinus rhythm
   * Significant QTc prolongation (≥ 480 ms)
   * New or previously unknown ischaemic changes that persist on repeat EKG:
   * ST elevations
   * T-wave inversions

   vi. Abnormal screening serum electrolytes and/or liver function tests

   vii. Laboratory evidence of prediabetic state or diabetes mellitus:
   * Hemoglobin A1c ≥ 5.7%, and/or
   * Fasting plasma glucose ≥ 100 mg/dL

   viii. Abnormal fasting lipids at screening (either of the following)
   * Triglycerides ≥ 150 mg/dL
   * LDL-cholesterol ≥ 160 mg/dL

   ix. Positive qualitative human chorionic gonadotropin beta subunit (β-hCG) (i.e., pregnancy test) in women of childbearing potential
3. COVID-19 precautions

   i. Unwillingness to comply with masking requirements per hospital policy

   ii. Active, documented COVID-19 at any time after screening through study completion
4. Reproductive concerns

   i. Women of childbearing potential not using highly effective contraception, defined as:
   * Surgical sterilization (e.g., bilateral tubal occlusion, bilateral oophorectomy and/or salpingectomy, hysterectomy)
   * Combined oral contraceptive pills taken daily, including during the study
   * Intrauterine device (levonorgestrel-eluting or copper) active at the time of the study
   * Medroxyprogesterone acetate (Depo-Provera®) injection active at the time of the study
   * Etonogestrel implants (e.g., Implanon®, etc.) active at the time of the study
   * Norelgestromin/ethinyl estradiol transdermal system (e.g., Ortho-Evra®) active at the time of the study

   ii. Women currently pregnant

   iii. Women currently breastfeeding
5. Any clinically relevant history or the presence of any active or chronic disease, including respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, etc. disease or diseases except for:

   * Osteoarthritis, not using chronic anti-inflammatory medications
   * Non-melanoma skin cancer, localized and not receiving systemic therapy
   * N.B. Minor chronic health problems that do not impair overall health/functional status and are judged unlikely to interfere with study conduct or data analysis may be permitted at the discretion of the PI
6. Currently taking any prescription medications other than vitamins or other nutritional supplements, subject to review by the PI

   o Any participant using biotin (vitamin B7) at >1000 international units per day must not take it for 3 d prior to any study blood draw due to interference with laboratory assays
7. Dermatologic concerns

   * History of cutaneous and/or mucosal eruptive reactions to food or drugs, including, but not limited to, rash or urticaria
   * Active skin conditions requiring ongoing care by a dermatologist except for localized non-melanoma skin cancer (not receiving systemic therapy)
8. Clinical concern for alcohol overuse at screening and/or by participant's report of consuming more than 14 standard drinks per week for males or more than 7 standard drinks per week for females
9. Current use of illicit drugs
10. Tobacco smoking currently or within the previous 6 months
11. History of or ongoing febrile illness within 30 days of screening
12. Any other disease or condition or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
13. Known allergy/hypersensitivity to any component of the medicinal product formulations (including soy or cow dairy), other biologics, venipuncture materials, plastics, adhesive or silicone, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
14. Dietary restrictions (e.g.., vegan, kosher, halal) on gelatin present in overencapsulation
15. Concurrent enrollment in another clinical study of any investigational drug therapy or use of any biologicals within 6 months prior to screening or within 5 half-lives of an investigational agent or biologic, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose | Day 4 (10 hours after dose)
  Fasting plasma glucose (units: mg/dL) after a single dose of alpelisib vs placebo.
Fasting serum insulin | Day 4 (10 hours after dose)
  Fasting serum insulin (units: micro-international units per milliliter, µIU/mL) levels after a single dose of alpelisib vs placebo.
Fasting serum C-peptide | Day 4 (10 hours after dose)
  Fasting serum C-peptide (units: ng/mL) after a single dose of alpelisib vs placebo.

SECONDARY OUTCOMES:
Overnight glucose profile | Days 3-4 (Approximately 24 hours)
  Glucose levels (units: mg/dL) serially sampled in interstitial fluid by continuous glucose monitor
Plasma glucose levels during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Measurement of plasma glucose levels (units: mg/dL) during OGTT in alpelisib vs placebo
Plasma glucose area under the curve (AUC) during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Plasma glucose AUC (units: arbitrary units) during OGTT in alpelisib vs placebo
Serum insulin levels during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Measurement of serum insulin levels (units: µIU/mL) during OGTT in alpelisib vs placebo
Serum insulin area under the curve (AUC) during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Serum insulin AUC (units: arbitrary units) during OGTT in alpelisib vs placebo
Serum triglyceride levels during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Measurement of serum triglyceride levels (units: mg/dL) during OGTT in alpelisib vs placebo
Serum free fatty acid levels during OGTT | Day 4 (Up to 180 minutes from the start of the procedure)
  Measurement of serum free fatty acid levels (units: mmol/L) during OGTT in alpelisib vs placebo
Fasting serum or plasma apolipoprotein B levels | Day 4 (10 hours after dose)
  Measurement of serum or plasma apolipoprotein B (units: mg/dL) in alpelisib vs placebo
Fasting serum total cholesterol levels | Day 4 (10 hours after dose)
  Measurement of fasting serum total cholesterol (units: mg/dL) in alpelisib vs placebo
Fasting serum high-density lipoprotein (HDL) cholesterol levels | Day 4 (10 hours after dose)
  Measurement of fasting serum HDL cholesterol (units: mg/dL) in alpelisib vs placebo
Fasting serum low-density lipoprotein (LDL) cholesterol levels | Day 4 (10 hours after dose)
  Measurement of fasting serum LDL cholesterol (units: mg/dL) in alpelisib vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Blood samples will be banked in our Insulin Resistance Biobank and will be made available to other researchers for legitimate research purposes upon request. Associated data will be shared along with specimens in the smallest possible quantity and on a need-to-know basis. No Protected Health Information (PHI) will ever be disclosed to other researchers. All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of an Institutional Review Board-approved Material Transfer Agreement (MTA) and/or Data Use Agreement (DUA), as appropriate.
Supporting Information: Study Protocol
Time Frame: Indefinitely following study completion.